CLINICAL TRIAL: NCT03598699
Title: A Multicenter, Vehicle-controlled, Randomized Study to Evaluate the Safety, Tolerability, Systemic Pharmacokinetics, and Pharmacodynamics of AXR-159 Ophthalmic Solution 3 mg/mL, 30 mg/mL, and 50 mg/mL in Patients With Dry Eye Disease (DED)
Brief Title: A Study to Evaluate AXR-159 Ophthalmic Solution in Patients With Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AxeroVision, Inc. (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AXR201701
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Results first posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-09

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AXR-159 Ophthalmic Solution 3 mg/mL (Experimental): AXR-159 Low Dose
  Interventions: Drug: AXR-159
- AXR-159 Ophthalmic Solution 30 mg/mL (Experimental): AXR-159 Mid Dose
  Interventions: Drug: AXR-159
- AXR-159 Ophthalmic Solution 50 mg/mL (Experimental): AXR-159 High Dose
  Interventions: Drug: AXR-159
- AXR-159 Ophthalmic Solution Vehicle (Placebo Comparator): Control Group
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: AXR-159 — AXR-159 Ophthalmic Solution
  Arms: AXR-159 Ophthalmic Solution 3 mg/mL; AXR-159 Ophthalmic Solution 30 mg/mL; AXR-159 Ophthalmic Solution 50 mg/mL
Drug: Vehicle — AXR-159 Ophthalmic Solution Vehicle
  Arms: AXR-159 Ophthalmic Solution Vehicle

SUMMARY:
Protocol AXR201701 is a multicenter, double-masked, vehicle-controlled, randomized, parallel group study carried out in 2 stages (Stage 1: AXR-159 Ophthalmic Solution (30 mg/mL or 50 mg/mL); Stage 2: AXR-159 Ophthalmic Solution (3 mg/mL, 30 mg/mL or 50 mg/mL) in approximately 430 patients diagnosed with dry eye disease (DED).

DETAILED DESCRIPTION:
Protocol AXR201701 is designed with 2 stages. For both Stages 1 and 2, patients with signs and symptoms of DED will be randomly assigned to receive either a single concentration of AXR-159 Ophthalmic Solution or AXR-159 Ophthalmic Solution Vehicle.

A screening visit will be followed by a baseline period where subjects will dose with AXR-159 Ophthalmic Solution Vehicle for 14 days. At the end of the baseline period patients who still exhibit signs and symptoms of DED will be enrolled into a 3-month double-masked treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older at screening visit
* Best-corrected visual acuity (BCVA) of 20/100 or better (Snellen equivalent), using the logarithm of the minimum angle of resolution (LogMAR) in each eye
* Reported history of dry eye for at least 6 months
* Corneal fluorescein staining score ≥ 2
* Eye dryness score ≥ 40
* Total Ocular Surface Disease Index (OSDI) score > 18

Exclusion Criteria:

* Uncontrolled ocular disease (except for dry eye disease/keratoconjunctivitis sicca) or uncontrolled systemic disease
* Patient has glaucoma, ocular hypertension, on IOP-lowering medications or have previously undergone any glaucoma laser or surgical procedure.
* Corneal abnormality or disorder that impacts normal spreading of the tear film (keratoconus, pterygia, scarring) or compromised corneal integrity
* BCVA worse than 20/100 in either eye
* Current use of punctal plugs, anticipated insertion during the study, or a history of punctal cautery in either eye
* Keratoconjunctivitis sicca secondary to destruction of conjunctival goblet cells
* Patients with clinically significant inflammation of the lid margin such as anterior blepharitis or ocular rosacea
* Recent (within the past 3 months) ocular surgery, trauma or herpes
* Use of contact lenses in either eye within one month prior to the screening visit or anticipated use during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-06-26 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2019-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail L Torkildson, MD, Principal Investigator — Andover Eye Associates, 138 Haverhill Street, Andover MA 01810; Kenneth R Kenyon, MD, Principal Investigator — Andover Eye Associates, 675 Paramount Drive, Raynham, MA 02767; Eugene McLaurin, MD, Principal Investigator — Total Eye Care, P.A., 6060 Primacy Parkway, Memphis, TN 38119
Locations (3):
- United States (3):
  - Andover Eye Associates, Andover, Massachusetts
  - Andover Eye Associates, Raynham, Massachusetts
  - Total Eye Care, P.A., Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited based on prespecified inclusion and exclusion criteria between June 2018 and September 2018. Of 265 subjects initially screened, 102 subjects were randomized. The first subject's screening visit was on June 26; the last subject's exit visit was on December 28.
Pre-assignment Details: All subjects who met the enrollment criteria at the initial screening visit were assigned to a 2-week run-in period on thrice daily topical vehicle. At the conclusion of the run-in period, 102 subjects again met the enrollment criteria and were randomized to either active or vehicle groups.
Groups:
- AXR-159 Ophthalmic Solution Vehicle: Control Group
  AXR-159: AXR-159 Ophthalmic Solution Vehicle
Period: Overall Study
Arm/Group | AXR-159 Ophthalmic Solution 50 mg/mL | AXR-159 Ophthalmic Solution Vehicle
Started | 54 | 48
Completed | 45 | 46
Not Completed | 9 | 2

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | AXR-159 Ophthalmic Solution 50 mg/mL | AXR-159 Ophthalmic Solution Vehicle | Total
Number analyzed (Participants) | 54 | 48 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.5 (10.72) | 65.3 (10.18) | 63.8 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 33 | 75
  Male | 12 | 15 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 51 | 47 | 98
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 47 | 39 | 86
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 54 | 48 | 102
Inferior Corneal Staining Score [Mean (Full Range); unit: units on a scale] — Score in the study eye based on Ora Calibra® Corneal and Conjunctival Staining Scale with a range from 0 to 4 (0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe). Higher numbers indicate more staining and a worse outcome. Population: Baseline Measure population = Modified Intent-to-Treat population with LOCF; Overall population = Safety population
  units on a scale
    number analyzed (Participants) | 50 | 47 | 97
    (all) | 2.16 [1.0 to 3.5] | 2.29 [1.0 to 4.0] | 2.22 [1.0 to 4.0]
Eye Dryness [Mean (Full Range); unit: units on a scale] — Using the visual analogue scale (VAS) subjects rated eye dryness on a subject level across both eyes by placing a vertical mark on the horizontal line to indicate the level of discomfort with a range of 0 to 100. 0% corresponds to "no dryness" (no discomfort) and 100% corresponds to "maximal dryness" indicating maximal discomfort. Population: Baseline Measure population = Modified Intent-to-Treat population with LOCF; Overall population = Safety population
  units on a scale
    number analyzed (Participants) | 50 | 47 | 97
    (all) | 76.8 [51 to 100] | 76.9 [48 to 100] | 76.9 [48 to 100]
Total Ocular Surface and Disease Index (OSDI) © for Dry Eye [Mean (Full Range); unit: units on a scale] — The 12-question OSDI © is assessed on a subject level on a total scale from 0 to 100, where higher scores represent greater disability. Population: Baseline Measure population = Modified Intent-to-Treat population with observed data only; Overall population = Safety population
  units on a scale
    number analyzed (Participants) | 50 | 47 | 97
    (all) | 50.9 [18 to 93] | 44.1 [18 to 98] | 47.6 [18 to 98]
Schirmer's Test [Mean (Full Range); unit: millimeters] — Unanesthetized Schirmer's Test measures the length of the moistened area of a test strip, placed in the lower temporal lid margin in the study eye, in mm following a 5-minute exposure period. Values of <10 mm are considered to represent a low tear volume. Population: Baseline Measure population = Modified Intent-to-Treat population with observed data only; Overall population = Safety population
  millimeters
    number analyzed (Participants) | 50 | 47 | 97
    (all) | 5.7 [1 to 10] | 6.4 [1 to 17] | 6.0 [1 to 17]
Tear Film Break-up Time (TBUT) [Mean (Full Range); unit: seconds] — Following the instillation of a sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye and several blinks over 30 seconds, the examiner monitored the integrity of the tear film with the aid of a slit lamp, noting the time it takes to form micelles from the time that the eye is opened. TBUT was measured in seconds using a stopwatch and a digital image recording system for the right eye followed by the left eye. Values reported are for the study eye. Population: Baseline Measure population = Modified Intent-to-Treat population with observed data only; Overall population = Safety population
  seconds
    number analyzed (Participants) | 50 | 47 | 97
    (all) | 2.239 [1.15 to 6.77] | 2.388 [0.82 to 5.46] | 2.311 [0.82 to 6.77]
Conjunctival Redness Score [Mean (Full Range); unit: units on a scale] — Assessed with the Ora Calibra® Conjunctival Redness Scale for Dry Eye. Scores range from 0 to 4 with 0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe; with higher numbers indicating more conjunctival redness. Values reported are for the study eye. Population: Baseline Measure population = Modified Intent-to-Treat population with observed data only; Overall population = Safety population
  units on a scale
    number analyzed (Participants) | 50 | 47 | 97
    (all) | 1.72 [1.0 to 3.0] | 1.61 [1.0 to 3.0] | 1.67 [1.0 to 3.0]
Total Lissamine Green Conjunctival Staining [Mean (Full Range); unit: units on a scale] — Change from baseline of Oxford Grading Scale measuring staining within a range from 0-5 (0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe, 5=Confluent) for each panel (temporal and nasal) and 0-10 as the sum of both panel scores for the total exposed inter-palpebral conjunctiva. Higher numbers indicate more staining and a worse condition. Values reported are for the study eye. Population: Baseline Measure population = Modified Intent-to-Treat population with observed data only; Overall population = Safety population
  units on a scale
    number analyzed (Participants) | 50 | 47 | 97
    (all) | 3.28 [0 to 8] | 2.96 [0 to 8] | 3.12 [0 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Inferior Corneal Staining Score
Description: Change from Baseline in Ora Calibra® Corneal and Conjunctival Staining Scale with a range from 0 to 4 (0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe) in the study eye. Higher negative scores mean a better outcome.
Time Frame: Month 3
Population: Modified Intent-to-Treat population with last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AXR-159 Ophthalmic Solution 50 mg/mL | AXR-159 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 50 | 47
units on a scale | -0.08 (0.65) | -0.03 (0.447)

2. Primary Outcome: Eye Dryness
Description: Change from baseline in Eye Dryness score on a subject level across both eyes. Using the visual analogue scale (VAS) subjects rated eye dryness by placing a vertical mark on the horizontal line to indicate the level of discomfort with a range of 0 to 100. 0% corresponds to "no dryness" (no discomfort) and 100% corresponds to "maximal dryness" indicating maximal discomfort. A greater negative change from baseline score means a better outcome.
Time Frame: Month 3
Population: Modified Intent-to-Treat population with last observation carried forward
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AXR-159 Ophthalmic Solution 50 mg/mL | AXR-159 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 50 | 47
units on a scale | -12.5 (22.62) | -14.9 (21.79)

3. Secondary Outcome: Total Ocular Surface and Disease Index (OSDI) © for Dry Eye
Description: Change from baseline in OSDI © score on a subject level. The 12-question OSDI © is assessed on a total scale from 0 to 100, where higher scores represent greater disability. A greater negative change from baseline indicates a better outcome.
Time Frame: Month 3
Population: Modified Intent-to-Treat with observed data only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AXR-159 Ophthalmic Solution 50 mg/mL | AXR-159 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 45 | 46
units on a scale | -8.8 (9.3) | -5.0 (16.93)

4. Secondary Outcome: Schirmer's Test
Description: Change from baseline in Schirmer's Test score in the study eye. Unanesthetized Schirmer's Test measures the length of the moistened area of a test strip, placed in the lower temporal lid margin of each eye, in mm following a 5-minute exposure period. Greater positive numbers indicate a better outcome.
Time Frame: Month 3
Population: Modified Intent-to-Treat population with observed data only
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | AXR-159 Ophthalmic Solution 50 mg/mL | AXR-159 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 45 | 46
millimeters | 0.8 (5.13) | 1.9 (6.77)

5. Secondary Outcome: Tear Film Break-up Time (TBUT)
Description: Change from baseline in the study eye with a greater positive increase indicating a better outcome. Following the instillation of a sodium fluorescein solution into the inferior conjunctival cul-de-sac of each eye and several blinks over 30 seconds, the examiner monitored the integrity of the tear film with the aid of a slit lamp, noting the time it takes to form micelles from the time that the eye is opened. TBUT was measured in seconds using a stopwatch and a digital image recording system for the right eye followed by the left eye. Values reported are for the study eye.
Time Frame: Month 3
Population: Modified Intent-to-Treat with observed data only
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | AXR-159 Ophthalmic Solution 50 mg/mL | AXR-159 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 45 | 46
seconds | -0.143 (1.093) | -0.178 (1.105)

6. Secondary Outcome: Conjunctival Redness Score
Description: Change from baseline of Ora Calibra® Conjunctival Redness Scale for Dry Eye. Scores range from 0 to 4 with 0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe; with higher numbers indicating more conjunctival redness. Greater negative numbers indicate a better outcome. Values reported are for the study eye.
Time Frame: Month 3
Population: Modified Intent-to-Treat population with observed data only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AXR-159 Ophthalmic Solution 50 mg/mL | AXR-159 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 45 | 45
units on a scale | 0.04 (0.673) | 0.26 (0.518)

7. Secondary Outcome: Total Lissamine Green Conjunctival Staining
Description: Change from baseline of Oxford Grading Scale measuring staining within a range from 0-5 (0=None, 1=Trace, 2=Mild, 3=Moderate, 4=Severe, 5=Confluent) for each panel (temporal and nasal) and 0-10 as the sum of both panel scores for the total exposed inter-palpebral conjunctiva. Larger negative numbers indicate reduced staining and a better outcome. Values reported are for the study eye.
Time Frame: Month 3
Population: Modified Intent-to-Treat population with observed data only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AXR-159 Ophthalmic Solution 50 mg/mL | AXR-159 Ophthalmic Solution Vehicle
Number analyzed (Participants) | 45 | 46
units on a scale | 0.40 (1.912) | 0.59 (1.758)

ADVERSE EVENTS:
Time Frame: For each subject, AEs were reported over a 12-week study period, starting from the randomization visit and start of treatment until the exit visit. Any serious adverse event (SAE) occurring during the study period and for 12 weeks after the last dose of study drug were to be immediately reported.
Description: All AEs spontaneously reported by the subject and/or in response to an open question from study personnel or revealed by observation, physical examination or other diagnostic procedures. Documentation as to the nature, date of onset, end date, severity, and relationship to Investigational Product, action(s) taken, seriousness, and outcome of any sign or symptom observed by the physician or reported by the subject upon indirect questioning.
Arm/Group | AXR-159 Ophthalmic Solution 50 mg/mL | AXR-159 Ophthalmic Solution Vehicle
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/54 | 1/48
Other Adverse Events (participants affected / at risk) | 34/54 | 7/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AXR-159 Ophthalmic Solution 50 mg/mL (N=54) | AXR-159 Ophthalmic Solution Vehicle (N=48)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Urethral Bleeding secondary to recent Cystoscope procedure; considered unrelated to study drug (vehicle) and resolved during study period
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AXR-159 Ophthalmic Solution 50 mg/mL (N=54) | AXR-159 Ophthalmic Solution Vehicle (N=48)
Dysgeusia (Nervous system disorders) | 20 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1
Instillation site pain (General disorders) | 9 | 2
Instillation site pruritus (General disorders) | 5 | 1
Eyelid oedema (Eye disorders) | 3 | 2
Eye pruritus (Eye disorders) | 3 | 1

LIMITATIONS AND CAVEATS:
The study was planned as a 2-stage study but has been terminated after completion of Stage 1 due to lack of funding.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
1. Master Clinical Development Agreement (MCDA) between AxeroVision and ORA stipulating written confidentiality agreement with third parties containing substantially similar restrictions on disclosure, use and other obligations contained in this MCDA.
2. Publication section in the Clinical Trial Protocol prohibiting individual publications without the company's consent.

DOCUMENTS (2):
  • Study Protocol (2018-02-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT03598699/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT03598699/SAP_001.pdf